CLINICAL TRIAL: NCT03859102
Title: Feasibility of Delivering Enhanced Recovery After Cardiac Surgery
Brief Title: Enhanced Recovery After Cardiac Surgery
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: James Cook University Hospital (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Principal Investigator, Dr Jim Coates, Clinical Research Fellow in Cardiothoracic Anaesthesia, James Cook University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRAS242926
Record Dates: First submitted 2018-12-28; First posted 2019-03-01 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Surgery; Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease; Tricuspid Valve Disease; Aortic Root Dilatation
Keywords: Enhanced recovery after Surgery; ERAS; Enhanced Recovery after Cardiac Surgery; Cardiac Surgery; Coronary Artery Bypass graft; Aortic Valve Surgery; Mitral Valve Surgery; Aortic Root Surgery
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease | interventions — Anesthesia, Local; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Sequential prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS Control/non-ERAS group (No Intervention): Standard usual care after cardiac surgery.
- ERAS group (Experimental): Enhanced Recovery After Cardiac Surgery. Pre-op carbohydrate drink, Lansoprazole and Gabapentin.
  Intra-operative: IV Paracetamol, Dexamethasone, Ondansetron, Local Anaesthetic to wounds.
  Post-op: Gabapentin PO, Paracetamol IV then PO, Ondansetron IV for 24hrs. Opiate sparing. Early extubation, early mobilisation, early removal of invasive devices. Early discharge.
  Interventions: Dietary Supplement: Pre-operative Carbohydrate PreLoad drink; Drug: Oral Gabapentin pre-op; Drug: Oral Lansoprazole pre-op; Drug: Intravenous Paracetamol intra-operatively; Drug: Intravenous Dexamethasone intra-operatively; Drug: Intravenous Ondansetron intra-operatively; Drug: Infiltration of surgical wounds with local anaesthetic; Drug: Intravenous Magnesium intra-operatively; Drug: Post-operative Gabapentin analgesia; Drug: Post-operative oral Paracetamol analgesia; Drug: Post-operative Ondansetron anti-emesis; Procedure: Early extubation; Procedure: Early mobilisation/physiotherapy; Other: Encourage early oral food intake

INTERVENTIONS:
Dietary Supplement: Pre-operative Carbohydrate PreLoad drink — Pre-operative Carbohydrate PreLoad drink, 1 sachet given the night before surgery. One sachet given 2-4hours before surgery.
  Arms: ERAS group
Drug: Oral Gabapentin pre-op — One dose of Gabapentin pre-operatively, 300mg orally.
  Arms: ERAS group
Drug: Oral Lansoprazole pre-op — One dose of Lansoprazole pre-operatively, 30mg orally.
  Arms: ERAS group
Drug: Intravenous Paracetamol intra-operatively — One dose of Paracetamol intra-operatively, 1gram intravenous infusion.
  Arms: ERAS group
Drug: Intravenous Dexamethasone intra-operatively — One dose of Dexamethasone intra-operatively as an anti-emetic, 8mg intravenous.
  Arms: ERAS group
Drug: Intravenous Ondansetron intra-operatively — One dose of Ondansetron intra-operatively as an anti-emetic, 4mg intravenous
  Arms: ERAS group
Drug: Infiltration of surgical wounds with local anaesthetic — Infiltration of surgical wounds with local anaesthetic at the end of surgery, Bupivacaine 1-2mg/kg.
  Arms: ERAS group
Drug: Intravenous Magnesium intra-operatively — One infusion of intravenous Magnesium Sulphate intra-operatively as an analgesic, 50mg/kg given over 30minutes.
  Arms: ERAS group
Drug: Post-operative Gabapentin analgesia — Post-operative oral Gabapentin 300mg, three times daily as an analgesic.
  Arms: ERAS group
Drug: Post-operative oral Paracetamol analgesia — Post-operative Paracetamol as an analgesic. Initially intravenously, then orally. One gram four times daily.
  Arms: ERAS group
Drug: Post-operative Ondansetron anti-emesis — Intravenous Ondansetron administered post-operatively as prophylactic anti-emesis. 4mg three times daily, for 24 hours. Then as required.
  Arms: ERAS group
Procedure: Early extubation — Removal of the endotracheal tube in the Intensive Care Unit as soon as is safe.
  Arms: ERAS group
Procedure: Early mobilisation/physiotherapy — Mobilisation (active and passive limb movements, deep breathing) with the assistance of nurse/physiotherapist to occur as soon as possible post-operatively.
  Arms: ERAS group
Other: Encourage early oral food intake — Patients will be encouraged to start eating as soon as possible post-operatively
  Arms: ERAS group

SUMMARY:
Enhanced Recovery Protocols (ERPs or bundles) have been established in many surgical specialties (such as colon cancer and orthopaedic joint surgeries) for several years in hospitals worldwide. The principles of Enhanced Recovery Protocols are those of early mobilization and restoration of normal function as soon as possible after surgery. These principles are achieved by use of alternate pain control regimens and removing invasive lines and drains as soon as possible. The benefits of ERPs are improved patient experience, earlier return to normal function and reduced length of stay. Enhanced recovery protocols for cardiac surgery have been published by the Enhanced Recovery After Cardiac Surgery Society.

The current study will investigate whether it is possible to utilise ERP bundles in the population of cardiac surgery patients at James Cook Hospital, with a view to rolling out a full ERP service. Secondary study outcomes will be patient-centred, including; pain scores, nausea and vomiting rates and time taken to return to normal function.

DETAILED DESCRIPTION:
Why? Enhanced Recovery Protocols (ERPs or bundles) have been established in many surgical specialties (such as colon cancer and orthopaedic joint surgeries) for several years in hospitals worldwide. The principles of Enhanced Recovery Protocols are those of early mobilization and restoration of normal function as soon as possible after surgery. These principles are achieved by use of alternate pain control regimens and removing invasive lines and drains as soon as possible. The benefits of ERPs are improved patient experience, earlier return to normal function and reduced length of stay. Enhanced recovery protocols for cardiac surgery have been published by the Enhanced Recovery After Cardiac Surgery Society. These protocols have been demonstrated as safe, though have yet to make it into mainstream practice in the UK. The use of ERPs in Cardiac Surgery has the potential to greatly improve the patient journey and hospital efficiency.

What? The current study will investigate whether it is possible to utilise ERP bundles in the population of cardiac surgery patients at James Cook Hospital, with a view to rolling out a full ERP service. Secondary study outcomes will be patient-centred, including; pain scores, nausea and vomiting rates and time taken to return to normal function.

Who? All adult patients over the age of 18 years and listed for cardiac surgery will be considered for inclusion in this study.

Where? The study population will be comprised of patients undergoing cardiac surgery at the James Cook University Hospital in Middlesbrough.

How? Study duration will be 6 months, with 80 patients (comprising a control and intervention group)

ELIGIBILITY:
Inclusion Criteria:

* Having Cardiac Surgery
* Aged 18 years or older at the time of consent
* Deemed appropriate for ERAS by Surgeon and Anaesthetist
* Able and willing to provide written informed consent

Exclusion Criteria:

* Aged 18 years or under
* Deemed not suitable for ERAS by Surgeon and/or Anaesthetist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-29 (Estimated)

PRIMARY OUTCOMES:
ERAS bundle compliance in the first 48hours post-op | 48hours post op
  Number of interventions for the ERAS protocol that are delivered to patient (numeric data e.g. 6 out of 10)

SECONDARY OUTCOMES:
Time to extubation | 0-24hours
  Time taken until patient extubated (ETT) post op (in minutes)
Time to mobilisation | 0-48hours
  First mobilisation with nurse/physiotherapist post-op (in minutes)
Time to oral diet | 0-48hours
  Time until patient first eats post-op (in minutes)
Post-op pain | 6hours
  Pain scores at 6hours, Numeric scale 0 (no pain) - 10 (severe pain)
Post-op pain | 12hours
  Pain scores at 12hours, Numeric scale 0 (no pain) - 10 (severe pain)
Post-op pain | 24hours
  Pain scores at 24hours, Numeric scale 0 (no pain) - 10 (severe pain)
Quality of Recovery | 6 weeks post surgery
  Quantification of patient quality of recovery. Using Q-o-R 15 Scale internationally validated scale. This allows the patient to report on a numerical scale from 0 (not at all) to 10 (all of the time); the patients scores on aspects of recovery such as pain at rest, pain on movement, quality of sleep, presence of nausea and vomiting, feeling supported by medical staff.

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Coates, MBBS, Principal Investigator — James Cook University Hospital
Locations (1):
- James Cook University Hospital, Middlesbrough, Teeside, United Kingdom

IPD SHARING:
Plan to Share IPD: No